CLINICAL TRIAL: NCT00942435
Title: A Randomized, Open Label Parallel Group Mechanical Prophylaxis Controlled Comparison Study With YM150, a Direct Factor Xa Inhibitor for Prevention of Venous Thromboembolism in Patients Undergoing Major Abdominal Surgery
Brief Title: A Study to Assess the Effect of YM150 for Prevention of Venous Thromboembolism in Patients Undergoing Major Abdominal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 150-CL-042
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Venous Thromboembolism
Keywords: YM150; Bleeding; VTE; FXa inhibitor; Deep Vein Thrombosis; Venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism; Hemorrhage; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- YM150 group (Experimental)
  Interventions: Drug: YM150
- mechanical prophylaxis group (Active Comparator)
  Interventions: Procedure: mechanical prophylaxis

INTERVENTIONS:
Drug: YM150 — oral
  Arms: YM150 group
Procedure: mechanical prophylaxis — The investigator will determine the method of mechanical prophylaxis
  Arms: mechanical prophylaxis group

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of the oral dose of YM150 for prevention of venous thromboembolism (VTE) in patients undergoing major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients after a major abdominal surgery
* Written informed consent obtained

Exclusion Criteria:

* Subject has history of symptomatic deep vein thrombosis and/or pulmonary embolism
* Subject has a hemorrhagic disorder and/or coagulation disorder
* Subject has had clinically important bleeding occurred within 90 days prior to the screening visit
* Subject has an active bacterial endocarditis
* Subject has uncontrolled severe or moderate hypertension, retinopathy, myocardial infarction or stroke
* Subject is receiving anticoagulants/antiplatelet agents
* Subject has a thrombocytopenia
* Body weight less than 40 kg at the screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Composite assessment of venous thromboembolism events and all causes of death | Until day 12

SECONDARY OUTCOMES:
Incidence of venous thromboembolism | Until day 28
Incidence of bleeding events | Until day 28
All cause mortality | Until day 28

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (6):
- Japan (6):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Shikoku

REFERENCES:
- [Derived] Sakon M, Nakamura M. Darexaban (YM150) prevents venous thromboembolism in Japanese patients undergoing major abdominal surgery: Phase III randomized, mechanical prophylaxis-controlled, open-label study. Thromb Res. 2012 Sep;130(3):e52-9. doi: 10.1016/j.thromres.2012.06.009. Epub 2012 Jul 2. PMID 22762942